CLINICAL TRIAL: NCT04586491
Title: The Effect of Oral Care Protocol on Prevention of Oral Mucositis in Pediatric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Dokuz Eylul University, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gülçin Özalp Gerçeker
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Mucositis; Pediatric Cancer; Oral Cavity
MeSH Terms: conditions — Mucositis; Neoplasms | interventions — CARE protocol; Mouthwashes; Solutions; Toothbrushing

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, parallel trial design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group/ Oral care protocol with saline solution (Experimental): All patients took oral care protocol in the unit with saline solution
  Interventions: Combination Product: Oral care protocol
- Control group/ Oral care protocol with sodium bicarbonate solution (Experimental): All patients took oral care protocol in the unit with sodium bicarbonate solution
  Interventions: Combination Product: Oral care protocol

INTERVENTIONS:
Combination Product: Oral care protocol — Oral care protocol
  Other Names: Daily evaluation of the inside of the mouth with the ChIMES; Gargle with solution; wiping the inside of the mouth with solution and sterile sponge; Brushing teeth with a soft toothbrush if platelet value was > 50000mm3.; Training for the child and family in oral care.

SUMMARY:
This study conducted to determine the effects of two oral care protocols containing sodium bicarbonate or saline solution in the prevention of oral mucositis (OM), mucositis degree, and recovery time in children with cancer.

DETAILED DESCRIPTION:
The study conducted as a randomized controlled trial with a parallel design with two groups; Study group/ Oral care protocol with saline solution Control group/ Oral care protocol with sodium bicarbonate solution

Study Hypothesis; There is a difference in oral mucositis (OM) between groups. There is a difference in the degree of OM between groups. There is a difference in the OM recovery time between groups. There is a difference in demographic variables in patients with and without mucositis.

The study sample was comprised of 43 children with cancer aged 1-17 years, received chemotherapy for ≥3 days at inpatient clinics, and whose families agreed to their participation in the study. Patients excluded who have oral ulceration or mucositis, taking any antiviral or antifungal therapy for OM before enrollment in the study. This trial was a triple blinded which the patients/parents, nurses, and the investigators have no idea about the groups.

In the study, patients were allocated by the blocked randomization. After naturally separating the gender variable into 2 layers, the age was divided into 5 layers as "<1 year, 1-3 years,>3-6 years, 6-12 years,>12 years", and the diagnosis variable was divided into 3 layers as "ALL, AML and oncological tumors."

Socio-Demographic Data Collection Form, International Child Mucositis Rating Scale (CHIMES), and Mucositis Follow-up Form used.

The child who do not have mucositis and who will be hospitalized for more than 3 days for chemotherapy will be distributed to the groups by stratified randomization method, the information of the patients will be obtained with the sociodemographic data collection form, oral care training will be given to the patient and the family, oral care protocol will be applied and it will be evaluated daily with the CHIMES and Mucositis Follow-up Form, and the severity of mucositis according to the World Health Organization Mucositis Assessment Index, the mean score of the CHIMES, recovery time will be monitored through the Mucositis Follow-up Form.

ELIGIBILITY:
Inclusion Criteria:

* have cancer, aged 1-17 years, received chemotherapy for ≥3 days at inpatient clinics and whose families agreed to their participation in the study.

Exclusion Criteria:

* who have oral ulceration or mucositis, in terminal period, taking any antiviral or antifungal therapy for OM before enrollment in the study.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
development of oral mucositis | until discharge from the hospital an average 1 week
  WHO Oral Mucositis Grading Scale: The WHO scale is dependent on both objective and subjective variables, and measures anatomical, symptomatic as well as functional components of oral mucositis.
  WHO Oral Mucositis Grading Scale

SECONDARY OUTCOMES:
severity of oral mucositis | until discharge from the hospital an average 1 week
  WHO Oral Mucositis Grading Scale: The WHO scale is dependent on both objective and subjective variables, and measures anatomical, symptomatic as well as functional components of oral mucositis.
  the Children's International Mucositis Evaluation Scale (ChIMES):It consists of seven elements: (1) Amount of mouth or throat pain(ChIMES1), (2) Effect of mouth or throat pain on swallowing(ChIMES2), (3) Effect of mouth or throat pain oneating (ChIMES3), (4) Effect of mouth or throat pain ondrinking (ChIMES4), (5) Receipt of pain medication (ChIMES5),(6) Receipt of pain medication for mouth or throat pain(ChIMES6), and (7) Presence of ulcers (ChIMES7).
recovery time of oral mucositis | until discharge from the hospital an average 1 week
  Mucositis Follow-up Form used for the recovery time

CONTACTS AND LOCATIONS:
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No